CLINICAL TRIAL: NCT05362656
Title: Preliminary Evaluation of the Artificial Intelligence Software VX1+ for the Detection and Automatic Tagging on 3D Mapping of Spatio-temporal Dispersion Areas During Atrial Fibrillation or Atrial Tachycardia Ablation Procedures.
Brief Title: AutoMatic disPERsion Tagging Function Preliminary Evaluation
Acronym: AMPERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Volta Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLIPL-03-001
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation; Atrial Tachycardia; Atrial Arrhythmia
Keywords: Artificial Intelligence; Cardiac ablation; Medical device; Software; Volta Medical; Atrial Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, non-randomized, non-controlled, single-center clinical investigation as part of the premarket clinical evaluation of VX1+ (medical device).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atrial mapping and dispersion auto-tagging with VX1+ (Experimental)
  Interventions: Device: VX1+ dispersion mapping

INTERVENTIONS:
Device: VX1+ dispersion mapping — Careful biatrial high density dispersion mapping is performed as the first step of the procedure. Operators map each region of both atria carefully by moving the mapping catheter slowly. If VX1+ application detects dispersion regions, the corresponding dipoles location will be automatically tagged on the 3D-map. Accuracy and relevance of dispersion regions should be confirmed by the operator by checking EGMs visually.

SUMMARY:
Interventional, prospective, non-randomized, single-center, non-controlled clinical investigation as part of the premarket clinical evaluation of VX1+ medical device, aiming to verify that VX1+ in bidirectional configuration with auto-tagging function is both ergonomic and reliable for dispersed electrograms detection and automatic tagging on 3D-map in real-time.

DETAILED DESCRIPTION:
Ablation of Atrial Fibrillation (AF) and Atrial Tachycardia (AT) is typically performed in predetermined anatomic regions of the left atrium (pulmonary veins isolation) and may be supplemented by a tailored ablation approach in order to identify areas of interest specific to the patient. The VX1+ medical device is intended to assist operators in the manual or automatic real-time annotation of 3D electroanatomical maps of the heart for the presence of multipolar intra-cardiac atrial electrograms exhibiting spatio-temporal dispersion during ablation procedures.

This study will specifically allow to evaluate the peroperative performance of VX1+ automatic tagging function in bi-directional configuration with a compatible 3D mapping system.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older.
* Patient candidate for catheter ablation of atrial tachycardia, or paroxysmal or persistent atrial fibrillation, de novo or after one or several previous ablation procedures.
* Continuous anticoagulation for more than 4 weeks before ablation.
* Patient giving his signed consent form to participate in the clinical study.
* Patient affiliated to the French social security

Exclusion Criteria:

* Contraindication to AF/AT catheter ablation.
* Major bleeding disorder.
* Contraindication to anticoagulation (Heparin, Warfarin or novel oral anticoagulants (NOAC)) or lack of anticoagulation for 4 weeks prior to the procedure.
* Presence of a left atrium (LA) thrombus on transesophageal echocardiography (TEE) prior to the procedure.
* Patient who is or could potentially be pregnant.
* Person deprived of liberty or under guardianship.
* Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-29 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Perioperative reliability of VX1+ in the real-time detection of electrograms in AF or AT exhibiting a spatio-temporal dispersion, and auto-tagging of these dispersion areas on 3D electroanatomical maps. | During procedure
  Comparison between the automatically annotated areas with VX1+ and those annotated manually following the operator's visual analysis (true positive, false positive, false negative).

SECONDARY OUTCOMES:
Accuracy of VX1+ in estimating cardiac cycle lengths | During procedure
  Comparison between the cardiac cycle length values estimated by VX1+ and the values measured manually by the operator from the electrograms signals (EGM).
Operators' satisfaction regarding the ergonomics of VX1+ | Through study completion, assessed up to 4 months
  Score of the operator's satisfaction and usage feedbacks regarding the ergonomics of VX1 +
Preliminary safety data on VX1+ perioperatively in terms of device deficiencies, adverse events and mapping time | From the date of hospitalization for the ablation procedure until the date of discharge, up to 1 week
  Rate of device deficiencies during the mapping phase, rate of Adverse Events for the hospitalization period and mapping time of dispersion areas with VX1+ device.

CONTACTS AND LOCATIONS:
Overall Officials: Julien SEITZ, MD, Principal Investigator — Hôpital Saint-Joseph Marseille
Locations (1):
- Hôpital Saint-Joseph, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seitz J, Bars C, Theodore G, Beurtheret S, Lellouche N, Bremondy M, Ferracci A, Faure J, Penaranda G, Yamazaki M, Avula UM, Curel L, Siame S, Berenfeld O, Pisapia A, Kalifa J. AF Ablation Guided by Spatiotemporal Electrogram Dispersion Without Pulmonary Vein Isolation: A Wholly Patient-Tailored Approach. J Am Coll Cardiol. 2017 Jan 24;69(3):303-321. doi: 10.1016/j.jacc.2016.10.065. PMID 28104073
- [Background] Seitz J, Durdez TM, Albenque JP, Pisapia A, Gitenay E, Durand C, Monteau J, Moubarak G, Theodore G, Lepillier A, Zhao A, Bremondy M, Maluski A, Cauchemez B, Combes S, Guyomar Y, Heuls S, Thomas O, Penaranda G, Siame S, Appetiti A, Milpied P, Bars C, Kalifa J. Artificial intelligence software standardizes electrogram-based ablation outcome for persistent atrial fibrillation. J Cardiovasc Electrophysiol. 2022 Nov;33(11):2250-2260. doi: 10.1111/jce.15657. Epub 2022 Sep 18. PMID 35989543
- [Result] Lotteau S, Seitz J, Bars C, et al. Bidirectional communication between an artificial intelligence device and a 3-dimensional navigation apparatus improves automation of multipolar electrogram mapping during paroxysmal and persistent atrial fibrillation. Cardiovascular Digital Health Journal. 2023;4(5):S8. doi:10.1016/j.cvdhj.2023.08.017